CLINICAL TRIAL: NCT06984978
Title: AI-assisted, Village Doctors and Express Services-Involved, Community-Based Multicenter Cluster Randomized Controlled Trial for Fall Prevention Among Rural Older Adults
Brief Title: EXpress Prevent Rural oldEr Adults' fallS, fractureS and Dependency (EXPRESS)
Acronym: EXPRESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yao Yao, Research professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20240805; 72374013 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-05-11; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Falls; Falls Injury; Fall Prevention
Keywords: AI-assisted fall prevention; Multicenter cluster randomized controlled trial; Fall-related injuries; Community-based intervention; Fall risks screening and assessment; Fall prevention; Rural older adults; Task shifting and sharing; Express

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted, village doctors and express services-involved personalized fall prevention strategy (Experimental): EXPRESS intervention is structured around five key components-SAFER.
  Interventions: Combination Product: AI-assisted, village doctors and express services-involved personalized fall prevention strategy
- Control group (No Intervention): The control group will receive standard health management through primary public health services and will be provided with a basic calendar to record fall events.

INTERVENTIONS:
Combination Product: AI-assisted, village doctors and express services-involved personalized fall prevention strategy — The EXPRESS trial implements a pragmatic, community-based, AI-assisted fall prevention strategy tailored to the needs of older adults in rural China. The intervention is structured around five core components-SAFER:
  1. Screening: multidimensional fall risk screening and assessment tailored to rural older adults;
  2. AI-assisted recommendations: AI-assisted personalized fall prevention recommendations;
  3. Fitness: Tailored balance and strength training via Health Intervention Cartoon Brochure and Action Demonstration Video;
  4. Events-based engagement: culturally integrated seasonal intervention packages following the traditional Chinese calendar;
  5. Reach-home delivery: home delivery of fall prevention services through local couriers.
  Arms: AI-assisted, village doctors and express services-involved personalized fall prevention strategy

SUMMARY:
Falls are the leading cause of injury-related death among individuals aged 65 and above in China. The incidence of falls shows a significant urban-rural disparity in China, with rural areas experiencing a markedly higher rate than urban regions. However, a systematic fall prevention strategy tailored to the needs of older people in rural China has not yet been established.

The EXPRESS study is a multicenter, cluster-randomized controlled trial designed to explore the effectiveness and health economic evaluation of an AI-assisted, village doctors and express services-involved, personalized fall screening and prevention strategy based on multidimensional risk profiling in reducing the incidence of falls and fall-related injuries among older people in rural China.

A total of 1,881 older individuals from 16 villages across four provinces in China (with four villages per province) will be recruited. These 16 rural areas will be randomly assigned to either the intervention group or the control group. The intervention group will receive the AI-assisted, village doctors and express services-involved personalized fall prevention strategy based on multidimensional fall risk screening and assessment, while the control group will follow routine primary health management practices.

The intervention period will last for one year, with randomization taking place after the baseline survey. The primary outcomes are the incidence of falls and fall-related injuries (including falls resulting in hospitalization and fractures, etc). Secondary outcomes include activity of daily living, quality of life, fall-related health literacy, depressive symptoms, cognitive function, dementia, physical function and performance, incidence of chronic non-communicable diseases, frailty, and sleep quality.

DETAILED DESCRIPTION:
The overall goal of EXPRESS is to develop an effective and sustainable fall prevention strategy suitable for rural China (AI-assisted, village doctors and express services-involved, personalized fall prevention strategy based on multidimensional risk profiling) to reduce the incidence of falls and fall-related injuries among older people in rural areas. The intervention strategy for the EXPRESS project is grounded in high-level evidence recommended by the guidelines, including the Technical Guidelines for Fall Prevention and Control in Community-Dwelling Older Adults published by China's National Health Commission. It aims to overcome the shortage of medical and human resources in rural China, leveraging social infrastructure to implement coherent interventions.

EXPRESS adopts a cluster-randomized multicenter design, recruiting older adults aged 65 and above from four provinces-Beijing, Hubei, Shanxi, and Anhui-selecting four villages from each province. The 16 villages are randomly assigned to the intervention or control group. The EXPRESS intervention is structured around five key components-SAFER, each designed to address rural health resource limitations, enhance accessibility, and provide personalized fall prevention services through AI technology and community integration.

S - Screening: Fall risk screening and assessment tailored to rural older adults. All participants undergo comprehensive fall risk assessments through a dual approach. First, village doctors administer a 10-item rural-adapted fall risk scale, developed by the research team for ease of use and specificity to the rural aging population. The scale captures key indicators such as mobility, balance, and prior fall history, offering a structured yet practical tool for frontline healthcare workers in resource-limited settings. Second, participants are instructed to complete sit-to-stand and 6-meter walking task (3 meters out and back) at their natural pace on a marked 3-meter mat. The smartphone is mounted on a specialized tripod on the opposite side, 2 meters from the endpoint of the mat, with a 30° downward angle to optimize the motion capture field of view. These recordings are analyzed using deep learning model and AI-powered motion analysis to extract five objective dimensions associated with fall risk: (1) balance (via sway and bilateral symmetry), (2) gait speed, (3) stride length, (4) trunk rotation (via turning motion), and (5) lower limb strength (via sit-to-stand movement). This combined subjective-objective assessment ensures accurate risk assessment and supports tailored interventions. Importantly, this risk screening and tailored health counseling process has been designed to be embedded within China's National Essential Public Health Service (EPHS) framework, particularly under the older adult health management program, which requires village doctors to conduct an annual physical examination for all residents aged 65 and above. As part of this initiative, the EXPRESS project incorporates the fall risk assessment and individualized consultation into the existing annual check-up workflow, allowing the service to be delivered efficiently during the routine health visit. To further support integration and incentivize adoption, the EXPRESS project offers a performance-based subsidy of RMB 6 per older adult to village doctors who complete both the fall risk screening and individualized counseling during the EPHS check-up. This approach not only promotes the institutionalization of fall prevention services, but also enhances sustainability and alignment with national health priorities in rural China.

A - AI-assisted recommendations: Personalized, AI-assisted falls prevention suggestions and health education. Collected assessment data are integrated into a decision-support system powered by artificial intelligence, which synthesizes evidence-based guidelines, expert consensus, and real-world data. The AI system generates personalized fall prevention plans tailored to each participant's risk profile and rural lifestyle. These plans assist village doctors in making informed, evidence-based decisions and provide actionable recommendations suitable for local implementation. Through the "1+1" transmission mechanism, village doctors conduct one-on-one risk assessments and explain the plan's key content, improving older people's health literacy and awareness of fall prevention. Meanwhile, a risk assessment and health recommendation report combining text and images will be issued to participants, using large fonts and including risk warning icons to ensure they are age and cultural appropriate.

F - Fitness: Tailored balance and strength training via Health Intervention Cartoon Brochure and Action Demonstration Video. Based on the risk assessment results, each older person will receive an individualized training recommendation customized by rehabilitation experts, which includes targeted training movements (such as balance training, lower limb strength training, etc.), supporting graphic and textual list (large font, easy to understand), and operation demonstration videos. Additionally, exercise rehabilitation experts develop a manual with 10 low-barrier exercises suitable for rural life scenarios, such as "bench balance training" and "big arm swings." Instructional videos are distributed to village doctors and participants. Village doctors are encouraged to lead group exercise sessions at village clinics, creating a community-driven atmosphere for physical activity.

E - Events-based engagement: Seasonal prevention activities and prevention materials integrated with traditional festivals and solar terms of the traditional Chinese calendar. To improve community engagement and intervention sustainability, the EXPRESS trial designed three round of intervention leveraging seasonal intervention packages that align with key traditional cultural events: the Chongyang Festival (October), the Spring Festival (January/February), and the Qingming Festival (April). These packages include culturally relevant and visually engaging materials, such as fall prevention calendars, fans printed with safety messages, and weather-specific tips. In addition, each package includes seasonal fall prevention tips, such as staying indoors during snowy weather, wearing non-slip shoes in winter, and being cautious during spring farming activities, thereby strengthening fall prevention awareness among older adults. The distribution of these packages aims to strengthen and consolidate the knowledge, beliefs, and behaviors of fall prevention among participants at different time points, leveraging local traditions to promote adherence, enhancing their sense of participation and sustainability in the intervention.

R - Reach-home delivery: The final and most important intervention strategy is home delivery of fall prevention services by express service. To alleviate the burden on village doctors and address the shortage of healthcare personnel in rural areas, the EXPRESS trial inspired by the Task Shifting/Sharing Theory and incorporates local couriers as community health support agents. Fall prevention intervention materials are remotely prepared by the technical team and distributed through a task-sharing platform. These couriers did their routine job and delivered intervention materials-including personalized health reports, educational calendars, and seasonal care packages-directly to participants' homes. This delivery model ensures the timeliness and coverage of fall prevention services to the doorsteps of older adults in rural and other regions with limited health care personnel.

The control group will receive standard health management through Primary Public Health Services and will be provided with a basic calendar to record fall events.

The intervention will last for one year, with participants being followed up on fall and injury incidents every three months. The primary outcome is the incidence of falls and fall-related injuries during the year of intervention. To reduce recall bias, fall and injury records will be collected using multiple methods: first, self-reporting by older adults on the calendar; second, a quarterly check-up by the couriers; and third, an endpoint assessment in the twelfth month of the study. Secondary outcomes include changes in activity of daily living, quality of life, fall-related health literacy, depressive symptoms, cognitive function, and dementia. The baseline data collection for this study was completed in August 2024, and the intervention effectiveness and health economic evaluation are expected to be completed by August 2025.

ELIGIBILITY:
Inclusion Criteria for Villages:

The village has a health clinic with at least one full-time village doctor.

Village officials and village doctors are actively cooperative and willing to participate in the study.

The village is located more than 2 kilometers away from other villages.

Exclusion Criteria for Villages:

Administrative villages where the township government is located (due to potential bias from centralized use of medical resources).

Villages that have previously conducted any form of fall-related knowledge promotion or intervention trials.

Inclusion Criteria for Participants:

Age 65 years or older.

Resides in the village for at least 12 months.

Provides informed consent and is willing to voluntarily participate.

Exclusion Criteria for Participants:

Suffering from major diseases such as cancer or stroke.

Disability.

Severe cognitive impairment.

Severe visual or perceptual impairments.

Any other condition preventing participation in the intervention.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1881 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Fall incidence within 12 months (rate of falls per person-year) | Months 3, 6, 9, 12 after baseline survey
  Defined as the number of falls divided by total person-time of observation. To minimize recall bias in fall measurement, three methods will be employed: self-recording by older adults or their family members on a calendar, quarterly in-person inquiries by delivery personnel, and final evaluation through interviews conducted by an assessment officer.
Proportion of participants with ≥1 fall within 12 months | Months 3, 6, 9, 12 after baseline survey
  A dichotomous outcome (fallers vs. non-fallers) that reflects risk reduction at the individual level. The measurement method is consistent with the fall incidence.
Fall-related injuries incidence within 12 months | Months 3, 6, 9, 12 after baseline survey
  Fall-related injuries included fractures, head injuries, hospitalizations, other events requiring medical attention. The measurement method is consistent with the fall incidence.

SECONDARY OUTCOMES:
Fall health literacy | Months 12 after baseline survey
  Fall health literacy as measured by a 15-item scale developed by the research team, with demonstrated reliability and validity. Each item is scored from 1 to 5, resulting in a total score ranging from 15 to 75. Higher scores indicate greater fall health literacy.
Activities of daily living | Months 12 after baseline survey
  Activities of daily living as measured by the Barthel Index. The Barthel Index total score ranges from 0 to 100, with higher scores indicating greater independence in daily activities.
Health-related Quality of life | Months 12 after baseline survey
  Health-related quality of life as measured by the EuroQol five-dimension five-level scale (EQ-5D-5L) summary index. The EQ-5D-5L index ranges from -0.391 to 1, with higher scores indicating better health status and quality of life.
Depressive symptoms | Months 12 after baseline survey
  Depressive symptoms as measured by the 5-item Geriatric Depression Scale (GDS-5). The GDS-5 total score ranges from 0 to 5, with higher scores indicating more severe depressive symptoms.
Cognitive function | Months 12 after baseline survey
  Cognitive function as measured by the Mini-Mental State Examination (MMSE). The MMSE total score ranges from 0 to 30, with higher scores indicating better cognitive function.
Dementia | Months 12 after baseline survey
  Dementia severity as measured by the Clinical Dementia Rating (CDR), evaluated by a professional physician. The CDR global score ranges from 0 (no dementia) to 3 (severe dementia), with higher scores indicating greater dementia severity.
Incidence of chronic non-communicable diseases | Months 12 after baseline survey
  The chronic non-communicable diseases include hypertension, diabetes, arthritis, sarcopenia, cervical spondylosis, heart problem, osteoporosis, kidney disease, hyperlipidemia, liver disease, lung disease, stomach disease, intestinal diseases. The incidence of chronic non-communicable diseases will be determined based on physician-diagnosed medical records, collected during routine health check-ups and follow-up visits by trained medical staff.
Frailty | Months 12 after baseline survey
  Frailty status as measured by the FRAIL scale. The FRAIL scale total score ranges from 0 to 5, with higher scores indicating greater frailty.
Sleep Quality | Months 12 after baseline survey
  Sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Gait Speed | Months 12 after baseline survey
  Gait speed as measured by the AI-assisted analysis of a 6-meter walk test on a 3-meter mat.
Stride Length | Months 12 after baseline survey
  Average stride length during the 6-meter walk test, assessed by AI-assisted video analysis.
Center of Pressure Sway Area | Months 12 after baseline survey
  Sway area of the center of pressure during a standardized standing or walking task, measured using AI-assisted video analysis.
Lower Limb Strength (Estimated Peak Force) | Months 12 after baseline survey
  Lower limb strength as measured by AI-assisted analysis of the sit-to-stand test, reported as estimated peak force.
Trunk Rotation Range | Months 12 after baseline survey
  Maximum trunk rotation angle measured during the 6-meter walk test, as assessed by AI-assisted video analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Yao, MD, Principal Investigator — Peking University
Locations (1):
- China Center for Health Development Studies, Peking University, Haidian, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Subject protection requirements

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT06984978/Prot_SAP_000.pdf